CLINICAL TRIAL: NCT04002544
Title: Topical Nitroglycerin to Facilitate Radial Arterial Catheter Insertion in Children: a Randomized Controlled Study
Brief Title: Nitroglycerin to Facilitate Radial Arterial Catheter Insertion in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: S72019
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Radial Artery Canulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NTG group (Active Comparator): In this group, nitroglycerin patch will be applied near the radial artery pulsation covered with a gauze.
  Interventions: Drug: NTG patch; Other: gauze cover
- Control group (Placebo Comparator): In this group, no patch as applied to the patient. However, a gauze will be applied to confirm blinding
  Interventions: Other: gauze cover

INTERVENTIONS:
Drug: NTG patch — A half-NTG patch (dose calculated at 5-12.5 mcg/kg/hr) will be applied to patients at the site of radial pulsation one hour before induction of anesthesia. The NTG patch will be applied to the right upper in half of the patients and will be applied to the left upper limb in the other half
  Arms: NTG group
Other: gauze cover — A gauze will be applied near the radial artery pulsation to ensure blinding

SUMMARY:
Local nitroglycerin (NTG) was successfully used as a vasodilator to facilitate cannulation of the radial artery. NTG was used in adults by topical application as well as subcutaneous infiltration. Subcutaneous infiltration of NTG resulted in significant vasodilatation, improved palpability of the radial artery, reduced the number of punctures and the time needed for cannulation in adults. Topical NTG was reported to increase radial artery diameter in healthy volunteers without reduction in arterial blood pressure. In pediatric population, there no sufficient evidence for the effectiveness of NTG in improving radial artery cannulation. In a case report on two neonates, topical nitroderm ointment successfully reversed tissue ischemia secondary to radial artery cannulation The aim of this work is to evaluate the use of topical NTG (patch) for increasing the diameter of radial artery, improving the cannulation success, and decreasing catheter-related ischemic complications.

DETAILED DESCRIPTION:
A written informed consent will be obtained from patient's parents or guardians. Randomization will be obtained using computer-generated sequence. Concealment will be obtained using opaque envelopes.

On arrival to the preparing room, patients will be randomized into one of the two groups:

- NTG group or, Control group

Ultrasound examination:

The diameter of radial artery will be measured using a linear, high frequency probe (12 mHz) of Simens machine. Measurement will be obtained in the short axis plane at the point with maximal pulsation. The point will be marked to guide the post-intervention examination. The operator will be an experienced single operator blinded to the study group. Measurements will be obtained in both limbs at baseline (before application of NTG patch application,30 minutes,60minutes after NTG application After induction of anesthesia, radial artery will be punctured by 22-g catheter by an experienced anesthetist

ELIGIBILITY:
Inclusion Criteria:

* children aged between 2 and 5 years scheduled for cardiac surgery

Exclusion Criteria:

* Systolic blood pressure less than 90 mmHg,
* previous radial artery puncture
* abnormal Allen's test
* hypercoagulable states
* coagulopathy
* previous vascular complications

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
change in The diameter of radial artery | 1 minutes before intervention then 30 and 60-minutes after the intervention
  mm

SECONDARY OUTCOMES:
palpability of radial pulse after NTG patch application | 1 minutes before intervention then 30 and 60-minutes after the intervention
  Grade 0: palpability did not change after NTG, grade 1: palpability improved after NTG, grade 2: palpability became bounding after NTG
Number of arterial punctures | 30 minutes
  number
successful cannulation confirmed | 30 minutes
  incidence
successful first-puncture cannulation | 30 minutes
  incidence
postoperative ischemic complications | 24 hours post intervention
  incidence
systolic blood pressure | 1 minute before the intervention, every 5 minutes for 1 hour
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Rady, Professor, Study Director — Head of department of anesthesia, Cairo University, Egypt
Locations (1):
- Ahmed Mohamed Hasanin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No